CLINICAL TRIAL: NCT01439438
Title: A Relative Bioavailability Study of Two Formulations of Topiramate 100 mg Coated Tablet in Healthy Male Volunteers, the Test Formulation Produced by Dr. Reddy's Laboratories Ltd. and the Reference Formulation (Topamax®) Marked by Janssen-Cilag Farmacêutica Ltda.
Brief Title: Topiramate Bioequivalence Study Brazil - Fast
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 116144
Record Dates: First submitted 2011-09-21; First posted 2011-09-23 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Epilepsy, Tonic-Clonic
MeSH Terms: conditions — Epilepsy, Tonic-Clonic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test formulation (Active Comparator): Test product: Topiramate 100 mg coated tablets produced by Dr. Reddy's Laboratories Ltd. in Period 1, followed by 28 days washout period during which no medication was administered; followed by reference product: Topamax® 100 mg coated tablets in Period 2
  Interventions: Drug: Topiramate coated tablet
- Reference formulation (Active Comparator): Topamax® 100 mg coated tablets marketed by Janssen-Cilag farmacêutica Ltda. in Period 1, followed by 28 days washout period during which no medication was administered; followed by test product: Topiramate 100 mg coated tablets produced by Dr. Reddy's Laboratories Ltd. in Period 2
  Interventions: Drug: Topamax® coated tablet

INTERVENTIONS:
Drug: Topiramate coated tablet — Test formulation
  Arms: Test formulation
Drug: Topamax® coated tablet — Reference formulation
  Arms: Reference formulation

SUMMARY:
This study is prospective, open-label, randomized, crossover, single dose, with 02 treatments, 02 sequences and 02 periods. The volunteers received, in each period, the reference or the test formulation, according to the randomization list, under fasting conditions, in order to evaluate if the reference and test formulations are bioequivalent.

DETAILED DESCRIPTION:
This study is prospective, open-label, randomized, crossover, single dose, with 02 treatments, 02 seuqences and 02 periods. The objective is to confirm if two formulations of topiramate 100 mg, coated tablet, are bioequivalent, after oral, single-dose administration under fasting conditions. The test product is topiramate 100 mg produced by Dr. Reddy's Laboratories Ltd. and the reference product is Topamax® marketed by Janssen-Cilag Farmacêutica Ltda. Twenty-eight healthy male volunteers were evaluated. The volunteers received, in each period, the test or the reference formulation, according to the randomization list. In each period, blood samples are collected in the following times: 00:00 (prior to the administration of medication); 00:20; 00:40; 01:00; 01:30; 02:00; 02:30; 03:00; 03:30; 04:00; 05:00; 06:00; 08:00; 12:00; 16:00; 20:00; 24:00; 48:00; 72:00; 96:00; 120:00; 144:00; 168:00; 192:00. The comparative bioavailability of the two formulations was evaluated based in statistical comparisons of relevant pharmacokinetic parameters, obtained from data of drug concentrations in blood.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 18 and 50 years
* Body mass index between 19 and 28,5 kg/m2
* Good health conditions
* Capable to understand the study's nature and aim, including risks and adverse effects and with intention to cooperate with the researcher and to act in compliance with requirements of the assay, this will be confirmed by the informed consent's signature

Exclusion Criteria:

* The volunteer has a known hypersensitivity to the study drug (topiramate) or to compounds chemically related
* History or presence of hepatic or gastrointestinal illnesses, or other condition that interferes over the drug's absorption, distribution, excretion or metabolism
* History of hepatic, renal, pulmonary, gastrointestinal, epileptic, hematologic or psychiatric illness; hypo or hypertension of any etiologic that needs pharmacologic treatment; has history or had myocardial infarction, angina and/or heart insufficiency
* Non-recommended electrocardiographic findings, according to investigator criteria, for the study's participation
* The results of the laboratory exams are out of the values considered as normal according to this protocol's rules, unless that they are considered as clinically irrelevant by the investigator
* The volunteer is a smoker
* The volunteer ingests more than 5 cups of coffee or tea a day
* Has history of alcohol or drugs abuse
* Use any regular drug within the 02 weeks that preceded the beginning of the treatment and the assessment date, or employed any drug that can interfere with the study within one week
* The volunteer was hospitalized for any reason within 08 weeks of the beginning of this study's first period of treatment and the assessment date
* Treatment within the 03 previous months of the study with any known drug that presents toxic potential for important organs
* The volunteer participated in any experimental study or ingested any experimental drug within the 06 months that precede the beginning of this study and the assessment date
* The volunteer donated or lost 450 mL or more of blood within the 03 months that preceded to the study initiation or donated more than 1500 mL within 12 months between the beginning of the study and the assessment date
* Consume of inductive drugs and/or enzymatic inhibitors (CYP450 - hepatic), that are toxic for the organism or presenting long half-life's elimination within the 04 weeks that precede the study's initiation
* Consume of alcohol in 48 hours antecedents to the admission to the study and along the study period
* Consume of food or beverages containing grapefruit (grapefruit) within 24 hours preceding each study period
* History of serious adverse reactions or hypersensitivity to any drug
* The volunteer has any condition that obstructs his participation in the study according the investigator's judgement

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2011-07-22 (Actual); Primary Completion 2011-09-11 (Actual); Study Completion 2011-09-11 (Actual)

PRIMARY OUTCOMES:
Area under curve of plasma concentration of drug from time 0 (zero) from time t (last measurable concentration) | Collection points from time 0 to 192 hours evaluated in two periods
  The area under the plot of plasma concentration of drug against time (non-compartimental method), after drug administration, defined as the area under the curve (AUC). The AUC 0-t is calculated from time 0 (prior to administration of medication) to time t (the time of the last quantifiable concentration), by linear trapezoidal rule. The AUC is of particular use in estimating the bioavailability of drugs, by measuring the extent of absorption.
Maximum observed concentration of drug through time (Cmax) | Collection points from time 0 to 192 hours evaluated in two periods
  Cmax is defined as the maximum or "peak" concentration of a drug observed after its administration. Cmax is one of the parameters of particular use in estimating the bioavailability of drugs, by measuring the total amount of drug absorbed. Measurement obtained directly of the plasma concentration curve of the drug (non-compartimental method). Occurring at Tmax.
Area under curve of plasma concentration of drug from the time 0 (zero) extrapolated to infinity (AUC0-inf) | Collection points from time 0 to 192 hours evaluated in two periods
  Measurement obtained directly from the plasma concentration curve of drug against time (non-compartimental method). AUC0-inf is calculated from time 0 (prior to administration of medication) extrapolated to infinity, by formula AUC0-inf=AUClast +Clast/Kel, where Clast is the Last measurable concentration and Kel is the first order rate constant associated with the terminal portion of the curve.
Time of maximum observed concentration (Tmax) | Collection points from time 0 to 192 hours evaluated in two periods
  Time when Cmax is obtained
Terminal half-life - T1/2 | Collection points from time 0 to 192 hours evaluated in two periods
  Calculated by formula: T1/2_Kel= Ln(2)/Kel.
First order rate constant associated with the terminal portion of the curve (Kel) | Collection points from time 0 to 192 hours evaluated in two periods
  This parameter is estimated by the angular coefficient of the regression line, calculated by the minimum squares method, of the natural logarithm of the concentration versus time for the last four concentrations values (or at least three) above the quantification limit

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Campinas, São Paulo, Brazil

REFERENCES:
- See also: Results for study 116144 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116144?search=study&search_terms=116144#rs